CLINICAL TRIAL: NCT07392606
Title: Assessment of Patient Experience in Telemedicine: Validation of the Co-designed "Patient Experience in Telehealth (PET)" Questionnaire to Measure Experience and Assess Environmental, Economic and Organizational Impact.
Brief Title: Validation of PET Questionnaire for Experience and Sustainability in Telemedicine. PET(Patient Experience in Telehealth)
Acronym: PET
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 8198
Record Dates: First submitted 2026-01-16; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: IBD; Arrythmia; Radiation Therapy Complication
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Telemedicine; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient Experience in Telehealth (PET) - questionnaire — The Patient Experience in Telehealth (PET) questionnaire was developed through a co-design process involving patients and healthcare professionals. The questionnaire includes a sociodemographic and telemedicine profile, followed by five Likert-scale sections covering access and technology use (6 items), communication with healthcare staff (5 items), privacy and safety (3 items), comfort, organization and integration of care (5 items), and economic and environmental impact (5 items). A general satisfaction section includes four items, plus one open-ended item for improvement suggestions. A supplementary in-depth section includes 11 items exploring avoided travel, time savings, caregiver involvement, device use, and interest in an automated carbon dioxide (CO₂) estimate. The questionnaire comprises 39 closed-ended items, 4 satisfaction items, 11 in-depth items, and 1 open-ended item. Completion time is approximately 10-15 minutes, and the survey is administered online in anonymous form.

SUMMARY:
Background: Telemedicine adoption has expanded rapidly in recent years, creating new opportunities for access to care, particularly for frail patients or those with mobility limitations. However, the large-scale deployment of remote healthcare services has highlighted the lack of validated instruments to systematically and multidimensionally assess patients' subjective experience. Patient experience is recognized as a key indicator of quality of care, with direct implications for treatment adherence, appropriate use of digital health technologies, and the effectiveness of organizational care models.

Rationale: No instruments have been specifically validated in Italy to measure patient experience in telemedicine. In response, the Fondazione Policlinico Universitario A. Gemelli - Istituto di Ricovero e Cura a Carattere Scientifico (FPG IRCCS) developed, through a co-design process involving expert patients and healthcare professionals, the Patient Experience in Telehealth questionnaire (PET). The tool was designed to capture not only overall satisfaction, but also relational, informational, and organizational domains, as well as perceived economic and environmental impact.

Objectives: The primary objective is psychometric validation of PET, assessing reliability and validity (construct, convergent, and discriminant). Secondary objectives include evaluating the perceived impact of telemedicine on care organization, patient-borne costs, and the environment, and exploring differences according to sociodemographic variables.

Methods: This cross-sectional observational study will administer PET to at least 200 adult patients who received one or more telemedicine services at FPG IRCCS within the preceding three months. Content validity will be assessed by an expert panel. Descriptive analyses, exploratory factor analysis (EFA), confirmatory factor analysis (CFA), and reliability testing will be performed. A subgroup will complete a test-retest assessment after 7-14 days.

Hypothesis: PET is expected to demonstrate satisfactory psychometric properties, discriminate across different levels of patient experience, and capture the perceived organizational, economic, and environmental impacts of telemedicine in healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Receipt of at least one telemedicine service at FPG IRCCS
* Provision of informed consent to participate in the study.

Exclusion Criteria:

* Cognitive or linguistic difficulties preventing comprehension of the questionnaire, in the absence of an available caregiver to provide assistance.
* Exclusive use of telemonitoring services or asynchronous reporting, as the survey focuses on synchronous interactions (e.g., video consultation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) who have received at least one telemedicine healthcare service at the Fondazione Policlinico Universitario A. Gemelli IRCCS (FPG IRCCS) across one or more specialist clinical areas. Participants will be consecutively recruited during the predefined data-collection period from among patients who received telemedicine services in the three months preceding study initiation, ensuring a heterogeneous sample with respect to age, sex, clinical condition, and level of digital familiarity.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Construct validity of the Patient Experience in Telehealth (PET) questionnaire | 1 month
  Construct validity of the PET questionnaire assessed through exploratory and confirmatory factor analysis.
Internal consistency and test-retest reliability of the Patient Experience in Telehealth (PET) questionnaire | 1 month
  Reliability of the PET questionnaire assessed by internal consistency and temporal stability.

SECONDARY OUTCOMES:
Overall satisfaction score measured by the Patient Experience in Telehealth (PET) questionnaire | 1 month
  Overall satisfaction with telemedicine services measured using a numeric rating scale included in the PET questionnaire. Score 0-10 (minimum 0, maximum 10)
Accessibility score measured by the Patient Experience in Telehealth (PET) questionnaire | 1 month
  Perceived accessibility of telemedicine services. Mean Likert-scale score (1-5)
Usability score measured by the Patient Experience in Telehealth (PET) questionnaire | 1 month
  Perceived ease of use of telemedicine technology. Mean Likert-scale score (1-5)
Perceived effectiveness score measured by the Patient Experience in Telehealth (PET) questionnaire | 1 month
  Perceived clinical effectiveness of telemedicine healthcare services. Mean Likert-scale score (1-5)
Organizational impact score measured by the Patient Experience in Telehealth (PET) questionnaire | 1 month
  Perceived impact on waiting times, care pathway simplification, and continuity of care. Mean Likert-scale score (1-5)
Patient-reported economic impact measured by the Patient Experience in Telehealth (PET) questionnaire | 1 month
  Perceived reduction in patient-borne costs, including travel expenses and avoided work leave. Likert-scale score (1-5) and self-reported avoided costs (€)
Patient-reported environmental impact measured by the Patient Experience in Telehealth (PET) questionnaire. | 1 month
  Perceived reduction in travel and associated environmental impact. Likert-scale score (1-5) and avoided travel distance (kilometers)
Association between PET domain scores and sociodemographic and clinical variables | 1 month
  Association between patient experience dimensions and participant characteristics, including age, educational level, and digital familiarity. Correlation coefficients and group comparisons

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Vetrugno, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS